CLINICAL TRIAL: NCT06127264
Title: Reliability of Force Measurement Within the Carbon Fiber Orthosis Proximal Cuff
Acronym: CuffForce
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Jason Wilken, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 202212359
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Ankle Foot Orthosis (AFO); Peripheral Neuropathy
Keywords: Ankle Foot Orthosis; Carbon Fiber Orthosis; Plantar Force
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Participants in Group 1 will be asked to fasten the proximal cuff to a self-selected cuff tightness 'SSCT', as well as three different predefined force levels; Loose, Moderate, and Tight. Participants in Group 2 and Group 3 will only be asked to fasten their AFO(s) to a self-selected tightness. Testing will occur without a CDO (NoCDO) and with each cuff tightness (SSCT, Loose, Moderate, Tight). Forces acting on the leg will be measured using wireless Loadpad sensors and forces acting on the plantar surface of the foot will be measured using wireless Loadsol insoles. Testing will include collection of force data as participants sit quietly, stand quietly, and walk and completion of questionnaires. Testing in the predetermined force levels (Loose, Moderate, Tight) will occur in a randomized order.
Who Masked: Participant
Masking Description: Participants will be blinded, to the greatest extent possible, to the different CDO proximal cuff tightness's.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- NoCDO (No Intervention): Participants will complete study activities without wearing a CDO
- SSCT (Experimental): Participants will complete study activities while wearing a CDO fastened to their self-selected proximal cuff tightness
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- Loose (Experimental): Participants will complete study activities while wearing a CDO fastened to a loose proximal cuff tightness
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- Moderate (Experimental): Participants will complete study activities while wearing a CDO fastened to a moderate proximal cuff tightness
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- Tight (Experimental): Participants will complete study activities while wearing a CDO fastened to a tight proximal cuff tightness
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)

INTERVENTIONS:
Device: Carbon Fiber Custom Dynamic Orthosis (CDO) — The carbon fiber custom dynamic orthosis (CDO) will consist of a semi-rigid carbon fiber footplate, a carbon fiber posterior strut, and a proximal cuff that wraps around the leg below the knee that is fastened to different tightness's
  Other Names: Ankle Foot Orthosis (AFO)
  Arms: Loose; Moderate; SSCT; Tight

SUMMARY:
The primary purpose of this research study is to determine if forces within carbon fiber custom dynamic orthoses (CDOs) can be reliability assessed using Loadpad and Loadsol force measuring sensors (Novel GMBH, St. Paul, MN). An improved understanding of the forces acting within orthoses may help to guide future orthosis related research studies, provision methods, and patient education.

Study participants will consist of three groups; 1) healthy, able-bodied adult participants using generic sized CDOs, which consist of a proximal cuff that wraps around the leg just below the knee, a posterior carbon fiber strut that runs the length of the leg and bends to store and return energy, and a semi-rigid footplate that acts as a lever arm to bend the posterior strut, 2) individuals without peripheral neuropathy who use AFO(s) regularly, and 3) individuals with peripheral neuropathy who use AFO(s) regularly. .

Group 1 participants will be asked to fasten the proximal cuff to a self-selected cuff tightness 'SSCT', as well as three different predefined force levels; 'Loose' where the proximal cuff is loosely fastened around the participants leg, 'Moderate' where the proximal cuff is fastened with moderate tightness, and 'Tight' where the proximal cuff is tightly fastened around the participants leg. Testing in the predetermined force levels (Loose, Moderate, Tight) will occur in a randomized order. Group 2 and Group 3 participants will be asked to fasten their AFO(s) to a self-selected 'SSCT' tightness.

For all groups, forces acting on the leg, within the proximal cuff, will be measured using wireless Loadpad sensors and forces acting on the foot will be measured using wireless Loadsol insoles. Testing will include collection of force data as participants sit quietly, stand quietly, and walk and completion of questionnaires.

DETAILED DESCRIPTION:
Ankle foot orthoses (AFOs) are medical devices often used to support the foot and ankle during daily activities. Carbon fiber custom dynamic orthoses (CDOs), one subset of AFOs, that consist of a proximal cuff that wraps around the leg just below the knee, a posterior carbon fiber strut that runs the length of the leg and bends to store and return energy during gait, a semi-rigid carbon fiber footplate that acts as a lever arm to bend the posterior strut, and in some cases a foam heel wedge placed between the footplate and the shoe. Different CDO design characteristics, such as posterior strut stiffness, device alignment, and heel cushion height and stiffness have been studied in the past. While different design characteristics have been studied previously, there is little information available concerning the proximal cuff and how it impacts patient outcomes. Different types of AFOs and CDOs have been used in an effort to offload the limb for years. Both CDOs and patellar tendon bearing (PTB) style AFOs have been shown to reduce forces acting on the plantar surface of the foot. While multiple studies have indicated the importance of fastening the proximal cuff, few have actually investigated the forces acting within the proximal cuff. A loose proximal cuff has been associated with pistoning of the limb, where the limb translates down within the proximal cuff during loading, potentially increasing forces acting on the foot and reducing the offloading effects of the orthosis. Only one study investigated the effects of altering forces within the proximal cuff by adding more padding to the proximal cuff, which was shown to improve limb offloading.

A better understanding of the forces acting within the proximal cuff, and how these effect patient outcomes would help to guide future AFO related research studies, provision, and patient education. At this point in time there is little guidance available to inform patients how tightly they need to secure the proximal cuff when wearing an AFO, many clinicians recommend tightening it so that it's secure, but not uncomfortable. The ability to measure forces within the proximal cuff and an idea of the range of forces seen in a clinical setting will act as a first step to better understanding how forces acting within the proximal cuff impact patient outcomes.

ELIGIBILITY:
Group 1 - Able Bodied Participants

Inclusion Criteria

* Between the ages of 18 and 65
* Healthy without current complaint of lower extremity pain, spine pain, open wounds or active infections, or medical or neuromusculoskeletal disorders that have limited their participation in work or exercise in the last 6 months
* Able to hop without pain
* Able to perform a full squat without pain
* Ability to read and write in English and provide written informed consent
* Ability to fit in a generic sized CDO

Exclusion Criteria

* Diagnosed with a moderate or severe brain injury
* Lower extremity injury resulting in surgery or limiting function for greater than 6 weeks
* Injuries that would limit performance in this study
* Diagnosed with a physical or psychological condition that would preclude functional testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
* Visual or hearing impairments that limit walking ability or limit the ability to comply with instructions given during testing
* Require use of an assistive device
* Unhealed wounds (cuts/abrasions) that would prevent AFO use
* BMI > 40
* Pregnancy

Group 2 - AFO Users without Peripheral Neuropathy

Inclusion Criteria:

* Between the ages of 18 and 90
* Use an AFO(s) for daily activities
* The AFO(s) proximal cuff is compatible with loadpad sensors
* Have used their AFO(s) for a minimum of 2 weeks
* Ability to walk 50 feet without use of an assistive device (e.g. cane, crutch, etc.)
* Ability to read and write in English and provide written informed consent

Exclusion Criteria

* Diagnosis or indication of peripheral neuropathy determined using Semmes Weinstein Filaments
* Medical or psychological condition that would preclude functional testing (ex. Moderate or severe brain injury, stroke, heart disease)
* Requirement of a knee stabilizing device (e.g. KAFO, KO) to preform daily activities
* Visual or hearing impairments that limit walking ability or limit the ability to comply with instructions given during testing
* BMI > 40
* Pregnancy

Group 3 - AFO Users with Peripheral Neuropathy

Inclusion Criteria:

* Between the ages of 18 and 90
* Use an AFO(s) for daily activities
* The AFO(s) proximal cuff is compatible with loadpad sensors
* Have used their AFO(s) for a minimum of 2 weeks
* Ability to walk 50 feet without use of an assistive device (e.g. cane, crutch, etc.)
* Diagnosis or indication of peripheral neuropathy determined using Semmes Weinstein Filaments
* Ability to read and write in English and provide written informed consent

Exclusion Criteria

* Medical or psychological condition that would preclude functional testing (ex. Moderate or severe brain injury, stroke, heart disease)
* Requirement of a knee stabilizing device (e.g. KAFO, KO) to preform daily activities
* Visual or hearing impairments that limit walking ability or limit the ability to comply with instructions given during testing
* BMI > 40
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proximal Cuff Force | Baseline
  Proximal cuff forces (N) will be measured as participants sit, stand, and walk without a CDO and in each CDO condition.
Peak Plantar Force | Baseline
  Plantar forces (N) will be measured across the total foot, the hindfoot, midfoot, and forefoot as participants sit, stand, and walk without a CDO and in each CDO condition.
Plantar Force Impulse | Baseline
  Plantar force impulse (Ns) across the total foot, the hindfoot, midfoot, and forefoot will be calculated using the integral of the force over the stance phase as participants sit, stand, and walk without a CDO and in each CDO condition.
Numerical Pain Rating Scale | Baseline
  Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable
Modified Socket Comfort Score (Comfort) | Baseline
  Comfort scores range from 0 = most uncomfortable to 10 = most comfortable

SECONDARY OUTCOMES:
Modified Socket Comfort Score (Smoothness) | Baseline
  Smoothness scores range from 0 = least smooth to 10 = most smooth

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wilken, PT,PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT06127264/Prot_SAP_000.pdf